CLINICAL TRIAL: NCT00465062
Title: A Study to Evaluate and Characterize the Effect of Pharmacological Chemicals on Blood From Patients With Gaucher Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070131; 07-N-0131
Record Dates: First submitted 2007-04-21; First posted 2007-04-24 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-03-03

CONDITIONS: Gaucher Disease
Keywords: Lysosomal Disease; Lipids; B Lymphocytes; Brain Damage; Gaucher Disease; GD
MeSH Terms: conditions — Gaucher Disease; Brain Injuries

SUMMARY:
Gaucher disease is a lysosomal storage disorder resulting from a deficiency in the key enzyme b-glucocerebrosidase (GCase). This enzyme is responsible for breaking down a specialized type of fat molecule, known as glucocerebroside, in the lysosome. The enzyme deficiency is caused by genetic mutations which result in the production of misfolded GCase protein. The absent or defective GCase enzyme activity leads to build-up of glucocerebroside inside certain cells. Over time, these Gaucher cells can accumulate and may cause inflammation or damage to specific areas within the body, including the liver, spleen, bone marrow, lung, and the central nervous system.

AT2101 is designed to act as a pharmacological chaperone by selectively binding to the misfolded GCase. After binding to the enzyme, it is thought that AT2101 promotes the proper folding, processing, and trafficking of the enzyme from the endoplasmic reticulum to its final destination, the lysosome, the area of the cell where the enzyme does its work. Once it reaches the lysosome, the pharmacological chaperone is displaced and the enzyme can perform its normal function, which is the breakdown of its natural substrate, glucocerebroside.

Several in vitro and in vivo preclinical studies have been conducted. In these studies AT2101 increased GCase enzyme level in cells derived from Gaucher disease patients with different genetic mutations, including cells with a genetic mutation associated with the neurologic form of Gaucher disease. In normal mice, oral administration of AT2101 resulted in a dose-dependent increase in GCase level in the liver, spleen, brain, and lung.

This study is designed to evaluate the ex vivo response to pharmacological chaperone therapy by testing blood samples from previously treated and untreated patients with Gaucher disease. The study will include patients with non-neuropathic Gaucher disease (type I) and neuropathic Gaucher disease (types II and/or III). Up to 50 patients will be enrolled at the NIH.

All subjects will participate in one study visit. Clinical information will be collected retrospectively from medical records. Information collected will include Gaucher disease diagnosis and history, medical history, family history, assessments of clinical severity, and genotype. A blood sample will be collected and various cells will be isolated for laboratory testing and research.

DETAILED DESCRIPTION:
Gaucher disease (GD) is a rare lysosomal storage disorder caused by mutations in the gene encoding acid-Beta-glucosidase (Beta-glucocerebrosidase [GCase]) (Gba), the lysosomal enzyme that catalyzes the breakdown of the lipid glucosylceramide (glucosylcerebroside [GlcCer]). The resulting deficiency in GCase activity leads to an intracellular accumulation of the substrate GlcCer, primarily in macrophage cells. These lipid-laden macrophages, known as Gaucher cells, are the hallmark of the disease and their accumulation in the liver, bone marrow, and spleen elicits the clinical symptoms associated with GD.

Pharmacological chaperone therapy is a novel approach to treat diseases due to protein misfolding/mistrafficking using small molecule ligands to rescue and increase the residual function of mutant proteins. For lysosomal storage diseases in which the causative mutant enzymes have residual activity, reversible inhibitors can act as pharmacological chaperones that specifically bind, stabilize, and facilitate the proper folding and trafficking of the mutant enzyme to the lysosome, thereby increasing its ability to degrade the accumulated substrate.

AT2101 (isofagomine [IFG] tartrate) is an iminosugar that functions as a selective pharmacological chaperone of GCase that is less stably folded as a result of missense mutations. Current data suggest that AT2101 may work by stabilizing mutant GCase in the endoplasmic reticulum and promoting trafficking of the enzyme to the lysosome. In the lysosome, when the pharmacological chaperone is displaced, the enzyme can perform its normal function, which is the breakdown of glucocerebroside.

This study is designed primarily to evaluate and characterize the effects of AT2101 on (GCase) activity and other markers of disease in lymphoblast and macrophage cell lines derived from patients with GD. Fifty subjects with a confirmed diagnosis of GD and a known Gba genotype will be enrolled in the trial.

The study will consist of one study visit. Clinical information will be collected retrospectively. Collected information will include but not be limited to GD diagnosis, medical history, family history, assessments of clinical severity and genotype. Blood samples for a series of ex vivo assays will be collected. Blood cell lines will be derived from the subjects' blood samples and used for the ex vivo assays, which will be conducted at a central laboratory.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for the study, subjects must fulfill all of the following inclusion criteria:

1. Willing and able to provide written informed consent by subject or legal guardian.
2. Male or female of any age.
3. Confirmed diagnosis of GD with known genotype.
4. Clinically stable and either treatment naive or on a stable dose of ERT and/or SRT for at least 6 months prior to study entry.
5. Available medical records for collection of retrospective clinical information.

EXCLUSION CRITERIA:

To be eligible for the study, subjects must not fulfill any of the following exclusion criteria:

1. Received any investigational product within 30 days prior to study entry.
2. Other significant disease or be otherwise unsuitable for the study, as determined by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2007-04-19; Study Completion 2008-03-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wong K, Sidransky E, Verma A, Mixon T, Sandberg GD, Wakefield LK, Morrison A, Lwin A, Colegial C, Allman JM, Schiffmann R. Neuropathology provides clues to the pathophysiology of Gaucher disease. Mol Genet Metab. 2004 Jul;82(3):192-207. doi: 10.1016/j.ymgme.2004.04.011. PMID 15234332